CLINICAL TRIAL: NCT01910064
Title: A Long Term Study of GK530G in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDT.07.SPR.27125
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GK530G (Experimental): GK530G is the fixed-dose combination gel of Adapalene and Benzoyl Peroxide, BPO
  Interventions: Drug: GK530G

INTERVENTIONS:
Drug: GK530G
  Other Names: Fixed-dose combination gel of Adapalene and Benzoyl Peroxide

SUMMARY:
This open label study is to determine the safety profile of GK530G in a long-term treatment (up to 12 months) in subjects with acne vulgaris and to evaluate the efficacy of GK530G in a long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at the age of 12 or older at the Screening visit.
* Those with clinical diagnosis of acne vulgaris with more than 20 non-inflammatory lesions (open and closed comedones) and 12 to 100 (inclusive) inflammatory lesions (papules, pustules and nodules) on the face (forehead, both cheeks, nose and chin).

Exclusion Criteria:

* Those with more than two nodular acne lesions or any cyst.
* Those with the diagnosis of any acne conglobata, any acne fulminans, any chloracne, or any drug induced acne.
* Those who have clinically significant abnormal findings or conditions on skin other than acne such as atopic dermatitis, perioral dermatitis, or rosacea that potentially interfere with study assessments according to Investigator's judgment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - Galderma investigational site, Urayasu, Chiba
  - Galderma investigational site, Fukuoka, Fukuoka
  - Galderma investigational site, Kawasaki, Kanagawa
  - Galderma investigational site, Yamato, Kanagawa
  - Galderma investigational site, Yokohama, Kanagawa
  - Galderma investigational site, Kumagaya, Saitama
  - Galderma investigational site, Chiyoda City, Tokyo
  - Galderma investigational site, Koto, Tokyo
  - Galderma investigational site, Machida, Tokyo
  - Galderma investigational site, Musashino, Tokyo
  - Galderma investigational site, Ōta-ku, Tokyo
  - Galderma investigational site, Shibuya City, Tokyo
  - Galderma investigational site, Shinjuku, Tokyo
  - Galderma investigational site, Suginami, Tokyo
  - Galderma investigational site, Tachikawa, Tokyo
  - Galderma investigational site, Kōtō City, Tpkyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 436 subjects have been enrolled in 20 site in Japan: First subject included: May 16, 2013; last subject out: July 18, 2014
Groups:
- GK530G: the fixed-dose combination gel of Adapalene and Benzoyl Peroxide
Period: Overall Study
Arm/Group | GK530G
Started | 436
Completed | 391
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | GK530G
Number analyzed (Participants) | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246
  Male | 190

OUTCOME MEASURES:

1. Primary Outcome: Local Tolerability (Erythema)
Description: Highest severity of Local tolerability scores worth than base line
Time Frame: 12 monhths
Measure: Number; unit: participants
Arm/Group | GK530G
Number analyzed (Participants) | 436
participants
  Mild | 149
  Moderate | 64
  Severe | 5

2. Primary Outcome: Local Tolerability (Scaling)
Description: Highest severity of Local tolerability scores worth than base line
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | GK530G
Number analyzed (Participants) | 436
participants
  Mild | 191
  Moderate | 60
  Severe | 2

3. Primary Outcome: Local Tolerability (Dryness)
Description: Highest Severity of Local Tolerability Scores Worse Than Baseline
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | GK530G
Number analyzed (Participants) | 436
participants
  Mild | 254
  Moderate | 52
  Severe | 1

4. Primary Outcome: Local Tolerability (Pruritus)
Description: Highest Severity of Local Tolerability Scores Worse Than Baseline
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | GK530G
Number analyzed (Participants) | 436
participants
  Mild | 149
  Moderate | 35
  Severe | 4

5. Primary Outcome: Local Tolerability (Stinging/Burning)
Description: Highest Severity of Local Tolerability Scores Worse Than Baseline
Time Frame: 12 months
Measure: Number; unit: subjects
Arm/Group | GK530G
Number analyzed (Participants) | 436
subjects
  Mild | 251
  Moderate | 79
  Severe | 9

6. Secondary Outcome: Percent Changes From Baseline in Total Lesion Counts
Time Frame: Baseline, Weeks 1, 2, 4, and Months 2, 3, 6, 9, 12
Measure: Median (Full Range); unit: percent change
Arm/Group | GK530G
Number analyzed (Participants) | 436
percent change
  Week 1 | 25.6 [-52 to 88]
  Week 2 | 42.1 [-87 to 93]
  Week 4 | 52.9 [-74 to 98]
  Month 2 | 67.1 [-65 to 100]
  Month 3 | 74.7 [-1 to 100]
  Month 6 | 82.0 [-81 to 100]
  Month 9 | 83.6 [-40 to 100]
  Month 12 | 86.2 [-16 to 100]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | GK530G
Serious Adverse Events (participants affected / at risk) | 6/436
Other Adverse Events (participants affected / at risk) | 311/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GK530G (N=436)
Peritonitis (Infections and infestations) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GK530G (N=436)
Nasopharyngitis (Infections and infestations) | 146 (199)
Gastroenteritis (Infections and infestations) | 17 (18)
Influenza (Infections and infestations) | 17 (17)
Skin irritation (Skin and subcutaneous tissue disorders) | 65 (73)
Pain of skin (Skin and subcutaneous tissue disorders) | 29 (30)
Eczema (Skin and subcutaneous tissue disorders) | 15 (19)
Dental caries (Gastrointestinal disorders) | 14 (15)
Headache (Nervous system disorders) | 18 (32)
Heat rash (Skin and subcutaneous tissue disorders) | 13 (14)
Dysmenorrhoea (Reproductive system and breast disorders) | 18 (79)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No